CLINICAL TRIAL: NCT00096603
Title: An Open Label, Multicenter Study to Evaluate the Safety of 1.0 mg/kg Subcutaneously Administered Efalizumab in Adults With Plaque Psoriasis Previously Enrolled in Study ACD2600g
Brief Title: A Study to Evaluate the Safety of Raptiva in Adults With Plaque Psoriasis Previously Enrolled in Study ACD2600g
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACD2601g
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Psoriasis
Keywords: Moderate to severe plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva (efalizumab)

SUMMARY:
This is an open label, multicenter study designed to evaluate the safety and tolerability of efalizumab administered subcutaneously at weekly doses of 1.0 mg/kg in subjects with plaque psoriasis who previously participated in Study ACD2600g.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Previous participation in Study ACD2600g
* For women of childbearing potential, continued use of an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to Efalizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2002-10; Study Completion 2004-07 (Actual)